CLINICAL TRIAL: NCT00435318
Title: Lateral Epicondylitis Iontophoresis Randomized Control Trial (LERCT)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study approval deferred by the IRB.
Sponsor: Vanderbilt University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 060984
Record Dates: First submitted 2007-02-12; First posted 2007-02-14 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Lateral Epicondylitis
MeSH Terms: conditions — Tennis Elbow | interventions — Iontophoresis

INTERVENTIONS:
Procedure: Iontophoresis

SUMMARY:
The intent of this double-blinded study is to investigate the short (2 months) and long-term (over 2 months) therapeutic capabilities of Iontophoresis.

DETAILED DESCRIPTION:
The intent of this double-blinded study is to investigate the short (2 months) and long-term (over 2 months) therapeutic capabilities of Iontophoresis. We anticipate that patients treated with Iontophoresis will have improved scores on the VAS and DASH assessments, and will recover more quickly than those patients receiving the Sham treatment. A Sham treatment is a method used in medical trials to help researchers determine the effectiveness of a drug/treatment which in this case will be Iontophoretic Administration using Dexamethasone. Placebos are inactive substances (Saline) used in this study to compare results with an active substance (Dexamethasone). Furthermore, it is the hope of this research team that through careful analysis and comparison of these two treatment arms a clear conclusion is met regarding the efficacy of Iontophoresis as a powerful treatment paradigm for patients suffering from this disorder.

ELIGIBILITY:
Inclusion Criteria

* Patients who have clinical evidence of Lateral Epicondylitis

  - Tests: Palpation of Lateral Epicondylitis, Resisted Wrist Extension, Middle Finger Test, Manual Muscle Test
* Patients who have symptoms (patient provided or documented information will be used to determine how long they have had symptoms) of Lateral Epicondylitis for at least a month, but no more than 3 months from most recent episode
* X-rays must show no evidence of post-traumatic or degenerative arthritis. All patients who present to VOI Hand & Upper Extremity Center complaining of Lateral Epicondylitis Symptoms have radiographs taken.

Patient selection factors include:

1. Ability and willingness to follow instructions
2. Patients who are able and willing to return for follow-up evaluations
3. Patients of all races and genders
4. Patients who are able to follow care instructions

Exclusion Criteria

* Patients less than 18 years old, or older than 75 years old
* Patients who to their knowledge our pregnant
* Patients unwillingly or unable to comply with a rehabilitation program, or who indicate difficulty or inability to return for follow-up visits prescribed by the study protocol
* Patients who qualify for inclusion in the study, but refuse consent to participate in the study
* Patients who have had non-steroidal anti-inflammatory drugs or systemic corticosteroids/analgesics within three days prior
* Patients who have local therapeutic modalities, such as: Iontophoresis, ultrasound, or heat within the last month
* Patients who have had:

  * Injection of steroids within the last year or prior surgery
  * Recurrent injury or previous fracture of affected area
  * History of Rheumatoid or Degenerative Arthritis, Carpal Tunnel Syndrome, Rotator Cuff abnormalities, neurologic abnormalities, muscular or shoulder dysfunction, peripheral neuropathy, radial nerve entrapment, fracture or tumor to the upper extremity, neck or thoracic pain, or pacemaker use.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-02; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Measuring using questionnaires and therapy measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Donald H Lee, M.D., Principal Investigator — Vanderbilt University